CLINICAL TRIAL: NCT03475550
Title: Managing Side Effects in Clinical Practice: A Quality Assurance Study in Functional Gastrointestinal Disorders
Brief Title: Managing Side Effects in Clinical Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Anthony Lembo, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017P000179
Record Dates: First submitted 2018-03-14; First posted 2018-03-23 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care 1 (Active Comparator): Patients will receive one of 2 different descriptions of the medication's risks and benefits. Both descriptions meet ethical standards of transparency and respect for person and are commonly used but have never been compared. "Standard of Care 1" includes more details than "Standard of Care 2".
  Interventions: Other: Standard of Care
- Standard of care 2 (Active Comparator): Patients will receive one of 2 different descriptions of the medication's risks and benefits. Both descriptions meet ethical standards of transparency and respect for person and are commonly used but have never been compared. "Standard of Care 2" includes fewer details than "Standard of Care 1".
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — The intervention involves clinician-provided information to patients receiving a new medication as part of their standard medical care. Intervention 1 includes more detailed information compared to Intervention 2.

SUMMARY:
This is a quality improvement health services study in the Division of Gastroenterology at Beth Israel Deaconess Medical Center (BIDMC).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate patients' reported experiences with regularly prescribed medications. No medications are prescribed as part of this study. Rather, if a patient are prescribed a new medication during their regularly scheduled clinic visit, he/she may be eligible to participate.

Patients who agree to participate and who are prescribed a medication in clinic will be contacted by telephone or email 3 weeks after their appointment to evaluate positive and negative experiences with the medication.

ELIGIBILITY:
Inclusion Criteria:

* Patient is seen in the Division of Gastroenterology at BIDMC
* Patient is prescribed a medication for the treatment of functional gastrointestinal disorders that has not previously been tried by the patient

Exclusion Criteria:

* Patient is not seen in the Division of Gastroenterology at BIDMC
* Patient has previously taken the drug that is prescribed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Patient-reported benefit from the drug | 3 weeks after the physician visit
  Visual Analog Scale of reported benefit from the drug (0-10)
Number of side effects reported from the drug | 3 weeks after the physician visit
  Checklist of reported side effects from the drug

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States